CLINICAL TRIAL: NCT00126360
Title: Pilot for a Randomised Comparison of Anastrozole Commenced Before and Continued During Adjuvant Radiotherapy for Breast Cancer Versus Anastrozole and Subsequent Ant-Oestrogen Therapy Delayed Until After Radiotherapy
Brief Title: STARS Breast Trial (Study of Anastrozole and Radiotherapy Sequencing Pilot)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St George Hospital, Australia (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STARS-Pilot (05/55 Graham)
Record Dates: First submitted 2005-08-02; First posted 2005-08-03 (Estimated); Last update posted 2005-11-10 (Estimated); Status verified 2005-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Timing of Radiotherapy; Local Control
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Drug: Timing of Anastrozole in respect to radiotherapy

SUMMARY:
This is a randomized study comparing the use of Anastrozole before and continuing during radiotherapy for breast cancer compared to the use of anastrozole after irradiation.

DETAILED DESCRIPTION:
Adjuvant radiotherapy is well established as the primary modality to enhance local control in breast cancer. The use of adjuvant hormone therapy such as tamoxifen has shown to improve local control to a relatively minor amount on its own and does enhance local control of adjuvant radiotherapy. There is however, conflicting in vitro and clinical data regarding the effects of different sequences on tamoxifen and radiotherapy in terms of both local control and enhancement of radiotherapy toxicities.

Aromatase inhibitors such as anastrazole are establishing themselves as a class of drug superior to tamoxifen for the control of estrogen dependent breast cancers and overall are better tolerated with the exception of greater bone loss.

As the key question is whether the sequencing of the aromatase inhibitor anastrozole alters local control by acting as an enhancer of the radiation breast cancer cell kill, it is therefore the aim of this study to compare 3 months of anastrozole prior to radiotherapy versus 3 months of anastrozole after radiotherapy with a specific objective of reducing the baseline ratio of in- field radiotherapy failure from 6% to 3%.This pilot study is preliminary to a planned long term study to investigate local failure.

For the pilot a period of 6 months with all contributing centres open will provide a good test of recruitment matching estimates. 100 patients will provide a good sample to compare to the 270 tamoxifen treated women in the breast boost study for quality of life. It will also provide a 95% CI on the proportion of complying women in the order of ± 5% if 85 to 90 % of women comply.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or more years. No upper limit.
* Post total mastectomy or lumpectomy. All planned surgery complete.
* Margins clear (no tumour contacting the inked margin)
* Tumour oestrogen or progesterone receptor positive
* Planned dose to irradiated volumes at least the biological equivalent of 45 Gy in 25 fractions or more.
* ECOG 0-2
* Patients post menopausal using same criteria as ATAC study.
* Written informed consent

Exclusion Criteria:

* Previous radiotherapy to the area to be treated.
* Previous invasive malignancy within 5 years of current breast cancer diagnosis with the exception of cervix in-situ or skin cancer other than melanoma.
* Patients with clinical evidence of metastatic disease.
* Previous hormonal breast therapy.
* Ongoing hormone replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-08; Study Completion 2016-05

PRIMARY OUTCOMES:
Local failure within irradiation volume

SECONDARY OUTCOMES:
Early quality of life
Lung fibrosis
Also demonstration of recruitment capacity at lead trial centres

CONTACTS AND LOCATIONS:
Overall Officials: Ass. Prof. Peter H Graham, MBBS FRANZCR, Principal Investigator — Cancer Care Centre, St George Hospital, Sydney
Locations (4):
- Australia (4):
  - Liverpool Hospital, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - Campbelltown Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland